CLINICAL TRIAL: NCT05631691
Title: Impact of School Based Intervention on Psychosocial Factors Associated With Trauma Among Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Nayyab Khurshid, Phd Student (Principal investigator), Fatima Jinnah Women University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FJWU
Record Dates: First submitted 2022-09-20; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Interventional Study
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: In this study, participants will be screened initially and then by randomization groups will be formed for intervention and comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): school students
  Interventions: Behavioral: Support for Students exposed to Trauma Program
- Comparison Group (No Intervention): school students

INTERVENTIONS:
Behavioral: Support for Students exposed to Trauma Program — Support for students exposed to trauma program (SSET) is a school-based intervention program for students who have been exposed to traumatic events and exhibit signs of post-traumatic stress disorder (PTSD). (Jaycox, Langley, & Dean, 2009; Jaycox, Langley, Stein et al., 2009). SSET is specifically designed for school teachers, school counsellors, and other non-clinical staff. SSET program is a series of 10 structured lessons designed to reduce post-traumatic and depressive symptoms and improve functioning in school children exposed to traumatic events. it includes psycho-education, relaxation, cognitive restructuring, social problems solving and behavioral exposure.
  Arms: Experimental Group

SUMMARY:
The present study is designed to identifying the post-traumatic stress symptoms in children experiencing some traumatic event and to adapt and apply school based intervention (Support for students exposed to trauma SSET) to students who shows the symptoms of post-traumatic stress disorder.

DETAILED DESCRIPTION:
Childhood trauma is a major mental health problem in recent era. Children who experienced sudden trauma have difficulty in learning, poor concentration in schools, and faced emotional and behavioral difficulties (Holt, Finkelhor, Kantor, 2007). Children who have been exposed to traumatic event are at a higher risk of developing psychopathology followed by trauma (Alisic et al.,2014). The present study is designed to identifying the post-traumatic stress symptoms in children experiencing some traumatic event and to adapt and apply school based intervention (Support for students exposed to trauma SSET) to students who shows the symptoms of post-traumatic stress disorder. This school based intervention (SSET) will provides a basis for how students can address overwhelming emotions, can deal with their daily life stressors and proactively learn to address unhelpful or maladaptive cognitions in positive way. This study will help to aware parents and teachers about mental health needs of children and adolescents.

ELIGIBILITY:
Inclusion Criteria of the study is:

* meets the cut off score on scale CATS (child and adolescent trauma screen).
* students availability for intervention phase
* age range 10-16 years

Exclusion Criteria:

* students above 16 years and below 10 years will not be included in the study.
* receiving any psychological/Mental health services or taking antidepressants
* Students whose primary problem is child abuse .

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in symptoms of PTSD, psychological distress, behavioral problems and increases resilience and social support of students who have some traumatic exposure | 6 to 8 week sessions
  The outcome of this study is to reduces the symptoms of PTSD and psychological distress in students who have some exposure to traumatic event and to increases participants social support and resilience. Participants will be assessed before and after intervention by standardized questionnaires: Child and Adolescent Trauma Screen questionnaire, Revised Children Anxiety and Depression scale, Strength and Difficulty questionnaire, Perceived Social Support Scale, and Youth Resilience Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan, Muzaffarabad, Azad Kashmir, Pakistan